CLINICAL TRIAL: NCT01421472
Title: A Randomized, Phase 2 Trial of Preoperative MM-121 With Paclitaxel in HER2-negative Breast Cancer
Brief Title: A Trial of Preoperative MM-121 With Paclitaxel in HER2-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-02-02-07 (ARD11918)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-03

CONDITIONS: ER Positive, Her2 Negative Breast Cancer Patients; Triple Negative Breast Cancer Patients
Keywords: Breast Cancer; Neoadjuvant; Her2 negative; Her2 non-overexpressing; Estrogen Receptor Positive; Triple Negative; MM-121; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — seribantumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MM-121 (SAR256212) + paclitaxel (Experimental): 2 week run-in of MM-121 followed by MM-121 + dosing of paclitaxel IV, followed by standard dosing of doxorubicin IV plus cyclophosphamide IV, followed by surgery.
  Interventions: Drug: MM-121; Drug: Paclitaxel
- Paclitaxel only (Active Comparator): Standard dosing of paclitaxel IV, followed by standard dosing of doxorubicin IV plus cyclophosphamide IV, followed by surgery.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: MM-121 — MM-121 IV at 40 mg/mg loading dose on Cycle 1, Week 1 followed by 20 mg/mg weekly for all subsequent doses
  Other Names: SAR256212
  Arms: MM-121 (SAR256212) + paclitaxel
Drug: Paclitaxel — Standard dosing of paclitaxel IV, followed by standard dosing of doxorubicin IV plus cyclophosphamide IV, followed by surgery.

SUMMARY:
To demonstrate whether addition of MM-121 to paclitaxel is more effective than treatment with paclitaxel alone, when administered as part of the neoadjuvant treatment in Her2 negative locally advanced operable breast cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, Phase II study of preoperative MM-121 with paclitaxel in HER2-negative breast cancer. Patients will be randomized to receive paclitaxel with or without MM-121 for 12 weeks followed by 4 cycles of doxorubicin plus cyclophosphamide and subsequent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of ER positive, HER2 negative invasive breast cancer (Group 1) or invasive triple-negative breast cancer (Group 2)
* Free of metastatic disease
* ≥ 18 years old
* Female
* Had no prior treatment for any cancer
* Eligible for treatment with paclitaxel, doxorubicin and cyclophosphamide

Exclusion Criteria:

* Have a history of severe allergic reactions to paclitaxel or other drugs formulated in Cremaphor® EL
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals
Locations (38):
- United States (38):
  - Universito of Birmingham atAlabama, Birmingham, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Arizona Oncology Associates, Tuscon, Arizona
  - Marin Cancer Center, Greenbrae, California
  - PMK Medical Group, Oxnard, California
  - Wilshire Oncology Medical Group, Rancho Cucamonga, California
  - Florida Cancer Research Institute, Plantation, Florida
  - Piedmont Healthcare, Altanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Georgia Cancer Specialists, Marietta, Georgia
  - University Of Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beaumont Health Systems, Royal Oak, Michigan
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - Northwest Cancer Specialists, Portland, Oregon
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Medical City, Dallas, Texas
  - Texas Oncology - Dallas, Dallas, Texas
  - Texas Oncology - Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - Texas Oncology -El Paso, El Paso, Texas
  - Texas Oncology - Garland, Garland, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology Plano East, Plano, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Puget Sound Cancer Center, Seattle, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- HR+: MM-121+ Paclitaxel: Hormone-receptor positive (HR+) sub-group randomized to receive:
  2 week run-in of MM-121 (20 mg/kg weekly IV infusion over 60 minutes following a 40 mg/kg loading dose), followed by 4 cycles of MM-121 (20 mg/kg weekly) + Paclitaxel (80 mg/kg IV infusion weekly over 60 minutes) for 12 weeks, followed by 4 cycles of doxorubicin and cyclophosphamide (8 weeks)
- HR+: Paclitaxel Only: Hormone-receptor positive (HR+) sub-group randomized to receive:
  Paclitaxel (80 mg/kg IV infusion weekly over 60 minutes) for 12 weeks followed by standard dosing of doxorubicin IV plus cyclophosphamide IV, followed by surgery.
- TN: MM-121 + Paclitaxel: Triple Negative (TN) patients randomized to receive:
  2 week run-in of MM-121 (20 mg/kg weekly IV infusion over 60 minutes following a 40 mg/kg loading dose), followed by 4 cycles of MM-121 (20 mg/kg weekly) + Paclitaxel (80 mg/kg IV infusion weekly over 60 minutes) for 12 weeks, followed by 4 cycles of doxorubicin and cyclophosphamide (8 weeks)
- TN: Paclitaxel: Triple negative (TN) patients randomized to receive:
  Paclitaxel (80 mg/kg IV infusion weekly over 60 minutes) for 12 weeks followed by standard dosing of doxorubicin IV plus cyclophosphamide IV, followed by surgery.
Period: Overall Study
Arm/Group | HR+: MM-121+ Paclitaxel | HR+: Paclitaxel Only | TN: MM-121 + Paclitaxel | TN: Paclitaxel
Started | 67 | 33 | 64 | 32
Completed | 67 | 33 | 64 | 32
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HR+: MM-121+ Paclitaxel | HR+: Paclitaxel Only | TN: MM-121 + Paclitaxel | TN: Paclitaxel | Total
Number analyzed (Participants) | 67 | 33 | 64 | 32 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.35) | 48.9 (10.53) | 49.3 (10.89) | 52.5 (13.45) | 50.25 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 33 | 64 | 32 | 196
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 13 | 3 | 36
  Not Hispanic or Latino | 57 | 22 | 51 | 29 | 159
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 7 | 4 | 11 | 5 | 27
  White | 57 | 26 | 48 | 26 | 157
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 5 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 67 | 33 | 64 | 32 | 196
Subject of Child-Bearing Potential (Y/N) [Number; unit: participants]
  Yes | 32 | 19 | 27 | 12 | 90
  No | 35 | 14 | 37 | 20 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR) (Rate of pCR)
Description: Pathologic Complete Response was defined as the absence of invasive cancer in the breast and lymph nodes following completion of neoadjuvant systemic therapy and reported according to the current AJCC staging system for neoadjuvant clinical studies. The endpoint was to determine the pathologic Complete Response (pCR) rates associated with weekly treatment of MM-121 plus paclitaxel followed by the combination treatment of doxorubicin plus cyclophosphamide compared with weekly paclitaxel alone followed by the combination treatment of doxorubicin plus cyclophosphamide in patients with human epidermal growth factor receptor 2 (HER2)-negative primary breast cancer.
Time Frame: At time of surgery, an expected average of 24-26 weeks
Population: Subjects with evaluable resection.
Measure: Number; unit: participants
Arm/Group | HR+: MM-121+ Paclitaxel | HR+: Paclitaxel Only | TN: MM-121 + Paclitaxel | TN: Paclitaxel
Number analyzed (Participants) | 66 | 30 | 56 | 29
participants
  Subjects with no pCR | 59 | 29 | 32 | 14
  Subjects with pCR | 7 | 1 | 24 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from a patient's first dose until 30 days after treatment termination. Serious adverse events were collected from time of informed consent until 30 days after treatment termination, or any time when assumed to be related
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination.
Arm/Group | HR+: MM-121+ Paclitaxel | HR+: Paclitaxel Only | TN: MM-121 + Paclitaxel | TN: Paclitaxel
Serious Adverse Events (participants affected / at risk) | 14/67 | 5/33 | 18/64 | 5/32
Other Adverse Events (participants affected / at risk) | 67/67 | 33/33 | 64/64 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HR+: MM-121+ Paclitaxel (N=67) | HR+: Paclitaxel Only (N=33) | TN: MM-121 + Paclitaxel (N=64) | TN: Paclitaxel (N=32)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 6 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 1 | 0
Breast Cellulutis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial Infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Infected Cyst (Infections and infestations) | 0 | 0 | 1 | 0
Infective Thrombosis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HR+: MM-121+ Paclitaxel (N=67) | HR+: Paclitaxel Only (N=33) | TN: MM-121 + Paclitaxel (N=64) | TN: Paclitaxel (N=32)
Nausea (Gastrointestinal disorders) | 52 | 24 | 48 | 24
Diarrhea (Gastrointestinal disorders) | 55 | 12 | 56 | 15
Constipation (Gastrointestinal disorders) | 12 | 13 | 27 | 15
Vomiting (Gastrointestinal disorders) | 16 | 10 | 17 | 7
Dyspepsia (Gastrointestinal disorders) | 13 | 8 | 18 | 8
Stomatitis (Gastrointestinal disorders) | 16 | 2 | 20 | 7
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 13 | 4 | 11 | 3
Abdominal Pain (Gastrointestinal disorders) | 7 | 4 | 10 | 2
Oral Pain (Gastrointestinal disorders) | 10 | 2 | 8 | 2
Hemorrhoids (Gastrointestinal disorders) | 6 | 0 | 9 | 2
Dry Mouth (Gastrointestinal disorders) | 5 | 3 | 2 | 2
Proctalgia (Gastrointestinal disorders) | 5 | 1 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Abdominal Distension (Gastrointestinal disorders) | 3 | 1 | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Mouth Ulceration (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 22 | 42 | 21
Rash (Skin and subcutaneous tissue disorders) | 28 | 5 | 27 | 8
Nail Disorder (Skin and subcutaneous tissue disorders) | 9 | 3 | 16 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 5 | 9 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 1 | 10 | 3
Nail Discoloration (Skin and subcutaneous tissue disorders) | 11 | 2 | 6 | 4
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 2 | 6 | 2
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 1 | 3 | 1
Skin Discoloration (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 2
Palmar-Plantar Erythrodysasthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 0 | 4 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 5 | 0 | 3 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 0
Nail Bed Tenderness (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 2
Dermatitis Acneform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Fatigue (General disorders) | 54 | 21 | 50 | 28
Mucosal Inflammation (General disorders) | 17 | 5 | 11 | 8
Pyrexia (General disorders) | 17 | 8 | 8 | 6
Peripheral edema (General disorders) | 10 | 9 | 11 | 6
Pain (General disorders) | 2 | 3 | 8 | 3
Asthenia (General disorders) | 3 | 2 | 4 | 2
Chills (General disorders) | 1 | 1 | 5 | 3
Chest Pain (General disorders) | 4 | 0 | 4 | 1
Catheter Site Pain (General disorders) | 0 | 2 | 3 | 1
Chest Discomfort (General disorders) | 2 | 2 | 1 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 2
Peripheral neuropathy (Nervous system disorders) | 32 | 17 | 37 | 18
Headache (Nervous system disorders) | 19 | 13 | 10 | 9
Dysgeusia (Nervous system disorders) | 14 | 8 | 20 | 5
Dizziness (Nervous system disorders) | 11 | 6 | 10 | 3
Peripheral sensory neuropathy9 (Nervous system disorders) | 8 | 5 | 9 | 2
Parasthesia (Nervous system disorders) | 7 | 4 | 6 | 4
Hypoasthesia (Nervous system disorders) | 2 | 2 | 5 | 3
Syncope (Nervous system disorders) | 4 | 1 | 2 | 1
Restless leg syndrome (Nervous system disorders) | 4 | 1 | 1 | 0
Hyperasthesia (Nervous system disorders) | 1 | 2 | 1 | 1
Sinus Headache (Nervous system disorders) | 0 | 0 | 2 | 3
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 4 | 11 | 4
Urinary Tract Infection (Infections and infestations) | 11 | 2 | 11 | 3
Sinusitis (Infections and infestations) | 5 | 0 | 6 | 2
Folliculitis (Infections and infestations) | 3 | 3 | 4 | 1
Oral Herpes (Infections and infestations) | 3 | 0 | 5 | 1
Oral Candidiasis (Infections and infestations) | 0 | 3 | 4 | 0
Fungal Infection (Infections and infestations) | 1 | 1 | 4 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 2 | 2
Nail Infection (Infections and infestations) | 3 | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 1 | 2 | 2 | 1
Candidiasis (Infections and infestations) | 2 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8 | 14 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 8 | 11 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 | 2 | 11 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 7 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 5
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 7 | 1 | 6 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 5 | 19 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 4 | 20 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 5 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 8 | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 2
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 2
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 18 | 7 | 17 | 11
Hypokalemia (Metabolism and nutrition disorders) | 21 | 3 | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 10 | 4 | 11 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 11 | 3 | 7 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1 | 7 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 1 | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 0 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 32 | 13 | 24 | 12
Neutropenia (Blood and lymphatic system disorders) | 21 | 9 | 18 | 7
Leukopenia (Blood and lymphatic system disorders) | 8 | 2 | 7 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 1 | 8 | 3
Leukocytosis (Blood and lymphatic system disorders) | 5 | 1 | 0 | 0
Weight Decreased (Investigations) | 19 | 5 | 17 | 8
Alanine Aminotransferase Increased (Investigations) | 5 | 2 | 4 | 0
Aspartate Aminotransferase Increased (Investigations) | 5 | 2 | 4 | 0
Insomnia (Psychiatric disorders) | 21 | 10 | 20 | 10
Anxiety (Psychiatric disorders) | 10 | 3 | 6 | 6
Depression (Psychiatric disorders) | 8 | 4 | 4 | 2
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 1
Hot Flush (Vascular disorders) | 10 | 6 | 8 | 8
Hypotension (Vascular disorders) | 6 | 2 | 5 | 2
Hypertension (Vascular disorders) | 2 | 3 | 3 | 0
Flushing (Vascular disorders) | 4 | 0 | 3 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 4 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 8 | 4 | 8 | 4
Dry Eye (Eye disorders) | 4 | 2 | 0 | 3
Lacrimatino Increased (Eye disorders) | 3 | 2 | 3 | 1
Conjunctivitis (Eye disorders) | 3 | 2 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 | 3 | 6 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 0
Breast Pain (Reproductive system and breast disorders) | 6 | 0 | 5 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 1 | 4 | 2
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 7 | 2 | 8 | 2
Pollakuria (Renal and urinary disorders) | 0 | 1 | 2 | 2
Urinary Incontinence (Renal and urinary disorders) | 2 | 1 | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 4 | 1 | 6 | 0
Palpitations (Cardiac disorders) | 4 | 1 | 3 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 2
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less